CLINICAL TRIAL: NCT04328818
Title: Indwelling Device-associated Biofilms in Oncological Critically Ill Patients
Brief Title: Indwelling Device-associated Biofilms
Acronym: BiofilmICU
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Olguta Lungu, Assistant lecturer, MD, Grigore T. Popa University of Medicine and Pharmacy
Other Study IDs: GTPopaUMPIASI
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Oncology; Critical Illness; Sepsis; Hospital Infection
Keywords: biofilm; oncologic; critical; Next Generation Sequencing
MeSH Terms: conditions — Neoplasms; Critical Illness; Sepsis; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples With DNA — Biofilm from four medical devices: endotracheal tube, arterial catheter, central venous catheter and urinary catheter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: indwelling device biofilm identification — performance of the NGS-based identification technique in comparison with the conventional culture-based one, for the same indwelling device biofilm sample

SUMMARY:
Healthcare associated infections linked to the use of indwelling medical devices increase hospital morbidity, mortality and the Intensive Care treatment costs. The essential strategy for mitigating these consequences are prompt source identifcation and control, with appropriate antimicrobial therapy initiation as soon as possible. Removing the source is one of the golden rule for infection control. Early identification of the responsible germs is the other major guiding element for the appropriate anti-infectious treatment.

Despite multiple detection/identification methods, there are no clear recommendations for biofilm identification in clinical practice. The gold standard method is bacterial/fungal culturing, with disadvantages related to late results, especially for slow growing, fastidious germs or related to the existence of uncultivable strains.

In order to obtain more sensitive, specific results and to increase the chances of better biofilm characterization, in the present study the investigators compare biofilm identification results obtained by standard cultivation methods with those by DNA amplification and next generation gene sequencing. The studied biofilm is associated to four criticallly ill oncological patients indwelling devices (endotracheal tube, central venous catheter, arterial catheter and urinary catheter).

DETAILED DESCRIPTION:
According to Regional Institute of Oncology, Iasi protocols, all septic patients with the need of invasive ventilatory support (endotracheal intubation), have concomitantly inserted a CVC, an AC and a UC, as standard of care. All patients undergo the protocol for the management of suspected/proven sepsis: initial resuscitation, specimen collection for microbiology/molecular biology tests, empirical/targeted anti-infectious treatment, source control, multiple organ support and treatment of the underlying disease/comorbidities. All RIO patients are screened for nasal, pharyngeal and rectal pathogen colonization at the time of hospital/ICU admission.

Informed consent - During the first 24 hours of ICU admission, all eligible patients will receive written information about the study: its implementation, aims, expected advantages and possible risks, and they will be asked to sign an informed consent. If the patient is unable to give consent at ICU admission due to pathological or drug-induced acute alteration of consciousness, a legal representative may give authorization. Once the participant regains the decision capacity, the individual will be asked to confirm or withdraw consent.

Swab sampling - The nasal, pharyngeal and rectal screening swab sampling is collected according to standard methods. In addition to this standard screening, in the first 24 hours of ICU admission cutaneous samples from the groin area of enrolled patients will be obtained, with sterile Copan eSwabTM swabs, a product recommended for aerobic, anaerobic and fastidious microbial agents.

Biofilm sampling and transport - The extraction of the four ID (ET, CVC, AC, UC) will be performed when the clinical condition of the patient dictates it (suspected catheter infection/no further need due to improvement or death). These devices will be extracted by medical ICU personnel, only at the indication and according to the medical judgment of the clinician, without being influenced by the patient's study participation.

Microbiological processing and analysis of the biofilm - Microbiological analysis will be performed by standard method: sample seeding on standard culture media, then biochemical identification test and AST according to CLSI standards and guidelines using MicroScan Walk Away 40 plus®, Beckmann Coulter automatic system compatible pannels.

Molecular biology processing and analysis of the biofilm - After complete sample collection, gene sequencing of the variable regions V3-V4 16S rRNA gene will be performed using Illumina MiSeq® Next Generation Sequencer System.

ELIGIBILITY:
Inclusion criteria:

1. Signed informed consent;
2. Age ≥18 years;
3. Suspected/proven sepsis/septic shock (Supplemental file 2);
4. APACHE II score ≥10 (Supplemental file 3);
5. Predictable invasive ventilatory support ≥ 48 hours;
6. Patient estimated survival ≥ 4 days.

Exclusion criteria:

1. Patient/legal representative refusal;
2. Age <18 years;
3. Chronic psychiatric/neurological disease with impaired decision-making capacity;
4. Pregnancy;
5. Invasive ventilatory support < 2 days;
6. Death in less than 4 days after ICU admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive critical oncology patients, which meet all inclusion criteria and have no exclusion criteria, admitted to the Intensive Care clinic of the Regional Oncology Institute, Iasi, Romania.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-06-05 (Actual); Primary Completion 2023-09-05 (Estimated); Study Completion 2025-10-05 (Estimated)

PRIMARY OUTCOMES:
The detection/identification of biofilm-associated pathogens | through study completion, an average of 1 year
  The detection/identification of biofilm-associated pathogens using Next Generation Sequencing (NGS) technique compared with standard microbiological diagnosis.

SECONDARY OUTCOMES:
Identification of pathogens involved in ID biofilm formation | through study completion, an average of 1 year
  Identification of pathogens involved in ID biofilm formation (ET, CVC, AC, UC) in the critically ill oncological patients.
Comparison of the biofilm-associated pathogens with those identified in currently used biological samples | through study completion, an average of 1 year
  Comparison of the biofilm-associated pathogens with those identified in currently used biological samples (tracheal aspirate/bronchoalveolar lavage, blood culture, urinary culture, surgical wound swab, etc.) collected from the same patient.
Comparison of the biofilm-associated pathogens with those identified in currently used biological samples (tracheal aspirate/bronchoalveolar lavage, blood culture, urinary culture, surgical wound swab, etc.) collected from the same patient. | through study completion, an average of 1 year
  Comparison of the biofilm-associated pathogens with those identified in currently used biological samples (tracheal aspirate/bronchoalveolar lavage, blood culture, urinary culture, surgical wound swab, etc.) collected from the same patient.
Establishing clinico-biological correlations | through study completion, an average of 1 year
  Correlations between biofilm-associated pathogens and patient clinico-biological data:
  * nasal, pharyngeal, rectal and skin pathogen screening;
  * associated risk factors: neutropenia, chemo/radiotherapy, corticosteroid treatment, previous anti-infectious therapy;
  * ID exposure time;
  * biological markers of inflammation;
  * diagnosed infection: respiratory tract infection, urinary tract infection, bloodstream infection, surgical site infection, sepsis of unknown origin, etc.;
  * severity scores: Sequential [Sepsis-Related] Organ Failure Assessment (SOFA) score, Acute Physiology and Chronic Health Evaluation II (APACHE II) score;
  * ICU and hospital LOS;
  * patient's outcome: survival/death;

CONTACTS AND LOCATIONS:
Overall Officials: Luminita Smaranda Iancu, Professor, Principal Investigator — University of Medicine and Pharmacy "Grigore T Popa", Iasi, Romania; Ioana Grigoras, Professor, Study Director — University of Medicine and Pharmacy "Grigore T Popa", Iasi, Romania; Olivia Simona Dorneanu, Assoc Prof, Study Director — University of Medicine and Pharmacy "Grigore T Popa", Iasi, Romania; Catalina Lunca, Assist Prof, Study Director — University of Medicine and Pharmacy "Grigore T Popa", Iasi, Romania; Teodora Vremera, Assist Prof, Study Chair — University of Medicine and Pharmacy "Grigore T Popa", Iasi, Romania; Stefania Brandusa Copacianu, MD, PhD, Study Chair — Regional Institute of Oncology, Iasi, Romania; Iuliu Ivanov, PhD, Study Chair — Regional Institute of Oncology, Iasi, Romania
Locations (1):
- Regional Institute of Oncology, Iași, Romania

IPD SHARING:
Plan to Share IPD: Undecided
Patient report form, patient microbiological study sheet, patient device study sheet.